CLINICAL TRIAL: NCT00036686
Title: A Clinical Trial of the Action of Isoflavones in Breast Neoplasia: Administration Prior to Mastectomy or Lumpectomy-A Pilot Study
Brief Title: Isoflavones in Treating Women Who Have Breast Cancer and Are Planning to Undergo Mastectomy or Lumpectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCC-13021; NCI-5348 (Other: NCI); NCI-P02-0214 (Other: NCI); 0104 (Other: CCOP)
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Soybean Proteins; Isoflavones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soy protein isolate (Experimental): Administration Prior to Mastectomy or Lumpectomy.
  Patients receive oral soy protein isolate twice daily and oral multivitamins once daily.
  Treatment continues for 2-4 weeks depending on time from study entry to planned surgical procedure.
  Interventions: Dietary Supplement: Soy protein isolate
- Placebo (Placebo Comparator): Administration Prior to Mastectomy or Lumpectomy.
  Patients receive oral placebo twice daily and oral multivitamins once daily.
  Treatment continues for 2-4 weeks depending on time from study entry to planned surgical procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Soy protein isolate — Arm I: Patients receive oral soy protein isolate twice daily and oral multivitamins once daily.
  Other Names: isoflavones
  Arms: Soy protein isolate
Other: Placebo — Arm II: Patients receive oral placebo twice daily and oral multivitamins once daily.
  Arms: Placebo

SUMMARY:
RATIONALE: Eating a diet rich in soy foods may slow the progression of some types of cancer. Isoflavones are compounds found in soy food that may slow the growth of breast cancer cells and prevent further development of breast cancer.

PURPOSE: Randomized pilot trial to study the effectiveness of isoflavones in preventing further development of breast cancer in women who are planning to undergo mastectomy or lumpectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of soy protein isolate (isoflavones) on modulation of intermediate endpoint biomarkers (such as cell proliferation, apoptosis, and steroid hormones) in women planning to undergo mastectomy or lumpectomy for breast cancer.
* Determine the effect of soy protein isolate on serum isoflavone levels in these patients.
* Correlate changes in serum isoflavones with changes in cell proliferation, apoptosis, and hormonal levels in patients treated with this therapy.
* Correlate the changes in cell proliferation and apoptosis with hormonal markers in patients treated with this therapy.

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are stratified according to the phase of the menstrual cycle at time of biopsy and time of surgery (follicular phase [i.e., during first 7 days of menstrual cycle] vs luteal phase [i.e., after day 7 of the menstrual cycle]). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral soy protein isolate twice daily and oral multivitamins once daily.
* Arm II:Patients receive oral placebo twice daily and oral multivitamins once daily.

In both arms, treatment continues for 2-4 weeks depending on time from study entry to planned surgical procedure.

PROJECTED ACCRUAL: A total of 106 patients (53 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing breast biopsy for any stage breast cancer

  * No excisional biopsy
  * At least one core biopsy block must contain carcinoma
* Definitive surgery (mastectomy or lumpectomy) planned for 2-4 weeks after registration to this study
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Premenopausal

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No known prior hepatic disease

Renal:

* No known prior renal disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective non-hormonal contraception
* No other prior malignancy except nonmelanoma skin cancer
* No known prior thyroid disease
* No adherence to vegan diet or other special dietary requirements that would preclude study participation
* No allergy to study agent
* No obesity (body mass index greater than 32)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent birth control pills or other hormonal therapy
* No concurrent thyroid hormone replacement medications

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* More than 30 days since prior antibiotics
* More than 4 weeks since prior soy products
* No routine consumption of greater than 40 mg of soy/day
* No other concurrent nutritional supplements, including modular supplements of other isoflavones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2002-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of Soy Protein Isolate Effect | 1 Year
  Determine the effect of soy protein isolate (isoflavones) on modulation of intermediate endpoint biomarkers (such as cell proliferation, apoptosis, and steroid hormones) in women planning to undergo mastectomy or lumpectomy for breast cancer.

SECONDARY OUTCOMES:
Occurrence of Effect on Serum Isoflavone Levels | 1 Year
  Determine the effect of soy protein isolate on serum isoflavone levels in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nagi B. Kumar, PhD, RD, FADA, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (7):
- United States (7):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Coastal Hematology and Oncology, P.C. - Savannah, Savannah, Georgia
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota